CLINICAL TRIAL: NCT02311309
Title: Epidemiology of Peroperative Bleeding and Transfusion During Scheduled Surgery.
Brief Title: Epidemiology of Severe Peroperative Bleeding During Scheduled Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: A13-D48-VOL.19
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Surgery; Blood Loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: Patients with either transfusion with pre ordered packed red blood cells or hemoglobin concentration > 8 g/dL.
  Interventions: Other: Control
- unanticipated bleeding: Unanticipated bleeding was defined as either transfusion above the pre ordered packed red blood cells or hemoglobin concentration < 8 g/dL.
  Interventions: Other: Unanticipated bleeding

INTERVENTIONS:
Other: Control — Control patients were defined as either transfusion using only pre ordered packed red blood cells or peroperative hemoglobin concentration >8 g/dL.
  Groups: control
Other: Unanticipated bleeding — Unanticipated bleeding was defined as either transfusion above the pre ordered packed red blood cells or peroperative hemoglobin concentration < 8 g/dL.
  Groups: unanticipated bleeding

SUMMARY:
Peroperative bleeding has been studied in specific populations exposed to bleeding (i.e. cardiac surgery, orthopedic surgery). Epidemiology of peroperative bleeding and transfusion remain poorly studied in the whole cohort of patients scheduled for surgery remain unknown. The investigators conducted a prospective study in order to examine the incidence, and risk factors associated with peroperative bleeding and transfusion.

DETAILED DESCRIPTION:
This was a prospective observational including all consecutive patients scheduled for surgery during a 3 month period.

Exclusion criteria were : emergency, cardiac surgery, and pediatric surgery. Patients received an oral information and informed consent was search for all of them.

Throughout the study period (3 months) data were prospectively recorded by members of a specific research team not involved in the care of patients. Preoperative, peroperative and immediate postoperative data (post anesthesia care unit) were collected.

Unanticipated bleeding was defined as either transfusion above the pre ordered packed red blood cells or hemoglobin concentration < 8 g/dL.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for non cardiac and non emergency surgery

Exclusion Criteria:

* Cardiac surgery
* Emergency surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients scheduled for surgery (expect cardiac, pediatric, and emergency surgery)
Sampling Method: Probability Sample
Enrollment: 1439 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Hanouz, M.D.,Ph.D., Principal Investigator — University Hospital, Caen

RESULTS

PARTICIPANT FLOW:
Groups:
- No Significant Bleeding: Patients in whom surgery did not resulted in significant bleeding
Period: Overall Study
Arm/Group | Control | Unanticipated Bleeding | No Significant Bleeding
Started | 541 (There were 863 patients with no peroperative bleeding in the 1439 patients studied) | 35 (There were 863 patients with no peroperative bleeding in the 1439 patients studied) | 863
Completed | 541 | 35 | 863
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Peroperative Significant Bleeding: Patients for whom surgery did not result in significant bleeding
- Total: Total of all reporting groups
Arm/Group | Control | Unanticipated Bleeding | No Peroperative Significant Bleeding | Total
Number analyzed (Participants) | 541 | 35 | 863 | 1439
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (17) | 66 (16) | 53 (19) | 56 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 19 | 405 | 678
  Male | 287 | 16 | 458 | 761
ASA class [Number; unit: participants] — ASA class reported in number of patients in a 4 class scale as defined by the American Society of anesthesiologists ASA 1 : otherwise healthy patient ASA 2 : A patient with mild systemic disease ASA 3 : A patient with severe systemic disease ASA 4 : A patient with severe systemic disease that is a constant threat to life
  participants
    ASA Class 1 | 107 | 2 | 261 | 370
    ASA Class 2 | 283 | 18 | 448 | 749
    ASA Class 3 | 150 | 14 | 150 | 314
    ASA Class 4 | 1 | 1 | 4 | 6
body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28 (6) | 27 (6) | 26 (6) | 27 (6)
red blood cell pre-planned (yes/no) [Number; unit: participants]
  Yes | 173 | 17 | 28 | 218
  No | 368 | 18 | 835 | 1221
Units of packed red blood cell pre planned (number) [Median (Inter-Quartile Range); unit: units of packed red blood cell] | 3 [2 to 3] | 3 [3 to 4] | 2 [2 to 3] | 3 [2 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Unanticipated Bleeding
Description: From arrival in operating room until the patients leave post anesthesia care unit
Time Frame: one day
Measure: Number; unit: percentage of participants
Arm/Group | Control | Unanticipated Bleeding | No Significant Bleeding
Number analyzed (Participants) | 541 | 35 | 863
percentage of participants | 0 | 100 | 0

2. Secondary Outcome: Transfusions
Description: transfusion pattern in the whole cohort
Time Frame: one day
Measure: Number; unit: number of participants
Arm/Group | Control | Unanticipated Bleeding | No Significant Bleeding
Number analyzed (Participants) | 541 | 35 | 863
number of participants
  transfusion of pack red blood cell | 33 | 31 | 1
  no transfusion | 508 | 4 | 862

3. Secondary Outcome: Preoperative Anemia
Description: proportion of patients with preoperative anemia
Time Frame: one day
Reporting Status: Not Posted

4. Secondary Outcome: Lowest Hemoglobin
Description: lowest peroperative hemoglobin concentration
Time Frame: one day
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control | Unanticipated Bleeding | No Peroperative Significant Bleeding
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes